CLINICAL TRIAL: NCT06868186
Title: A Multicenter, Randomized, Parallel-group Study to Evaluate Efficacy of Surgical Navigation System 'RUS NE' in Patient Underwent Robot-assisted Partial Nephrectomy
Brief Title: A Multicenter Study of RUS NE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hutom Corp (Industry)
Collaborators: Asan Medical Center (Other); Seoul National University Hospital (Other); Samsung Medical Center (Other); Chonnam National University Hospital (Other); Kyungpook National University Hospital (Other); Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTK-001
Record Dates: First submitted 2025-02-28; First posted 2025-03-10 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Renal Tumors
Keywords: renal tumor; robot assisted partial nephrectomy; 3D model; surgical navigation
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Experimental group will undergo robot-assisted partial nephrectomy for renal tumor using RUS NE.
  Interventions: Device: RUS NE
- Control arm (No Intervention): Experimental group will undergo robot-assisted partial nephrectomy for renal tumor without using RUS NE.

INTERVENTIONS:
Device: RUS NE — The RUS NE is an endoscopic imaging treatment planning software program. It creates a patient-specific simulation of the intra-abdominal surgical environments, allowing for the visualization of tumor, vascular structures and intra-abdominal organs during the surgical planning process and the operation. RUS NE utilizes preoperative CT images of the patients to segment tumor, organs, and blood vessels and reconstructs them into a 3D model. Although there is no direct intervention on the patient, the surgeon uses RUS NE as a surgical navigation tool to simulate the surgery before performing the actual procedure.
  Arms: Experimental Group

SUMMARY:
This sponsor-initiated, randomized controlled clinical trial aims to demonstrate the clinical efficacy of RUS NE Surgical Navigation System in patients undergoing robotic-assisted partial nephrectomy. The trial will compare the experimental group (n=102) using RUS NE with a control group (n=102), aiming to show an 10% reduction in operation time. The study will involve 6 medical centers in South Korea in patient recruitment and evaluate the clinical efficacy and feasibility of the software, which has been shown to be reliable in previous studies.

* Investigational Medical Device: RUS NE (Endoscopic Imaging Treatment Planning Software)
* Clinical Trial duration: 24 months from IRB approval -Target number of subjects: Total of 204 participants

DETAILED DESCRIPTION:
After selecting subjects and obtaining informed consent, randomization will be conducted. Robot-assisted partial nephrectomy will be performed using RUS NE or without using software. Parameters-associated with operation or clinical outcomes will be evaluated during hospitalization period or through outpatient follow-ups for up to 3 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were diagnosed with renal tumor and undergo robot-assisted partial nephrectomy
* The diameter of renal tumor is 7cm or below
* Individuals aged between 19 and 80
* Individuals who, before participating in the clinical trial, undergo an interview in a separate place, understand sufficient explanation of the purpose and content of the trial, and voluntarily sign informed consent form

Exclusion Criteria:

* Individuals with solitary kidney or horseshoe kidney
* Individuals undergo bilateral nephrectomy
* Individuals undergo operation other than partial nephrecotmy
* Individuals with a history of abdominal surgery and are expected to have severe intra-abdominal adhesion influencing the surgical outcomes
* Individuals with severe chronic kidney disease (eGFR < 45, calculated with EPI-CKI equation)
* Individuals with American society of anesthesiologists physical status classification (ASA) IV-VI
* Individuals with a history of psychosis, alcohol abuse or are expected not to adhere to the schedule of the clinical study
* Individuals who were participated in other clinical study within 4 weeks of screening
* Individuals who are thought to be inappropriate to participate to the clinical trial by the investigators

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Operative time | The operative day (operative day ± 5 days)
  The duration of time between starting a surgical incision to the last sutures of the operation.

SECONDARY OUTCOMES:
Tumor and vessel identification time | The operative day (operative day ± 5 days)
  The duration of time between starting manipulation of the surgeon console to the finishing dissection of the hilum and perinephric fat
Resection volume | From the postoperative 1week to the postoperative 5 weeks
  Calculated from the 3-dimensional lengths from the resected renal specimen using ellipsoid formula (π/6XYZ)
Postoperative complications | From the postoperative 8 weeks to the postoperative 16 weeks
  Incidence of postoperative complications occurred within 4 weeks after the operation. The complications include urine leak, acute kidney injury, renal hemorrhage, fluid collection, abscess, and pulmonary or cardiac complications.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryn Song, M.D.,Ph.D., Principal Investigator — Asan Medical Center
Locations (4):
- South Korea (4):
  - Chonnam National University Hospital, Kwangju, Jeollanam-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee S, Lee HY, Song C. Assessment of Feasibility and Outcomes of RUS Surgical Navigation System During Robot-Assisted Partial Nephrectomy for Small Renal Masses. Int J Urol. 2025 May;32(5):576-583. doi: 10.1111/iju.70014. Epub 2025 Feb 13. PMID 39945060